CLINICAL TRIAL: NCT03677349
Title: Evaluation of the Interest of the Neurorrhaphy in the Resensitisation of Free Flaps in Maxillofacial Reconstructive Surgery. Randomized Prospective Study.
Brief Title: Evaluation of the Interest of the Neurorrhaphy in Resensitizing Free Flaps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Hospital of Aurillac (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-392; 2017-A03470-53 (Other: 2017-A03470-53)
Record Dates: First submitted 2018-06-04; First posted 2018-09-19 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Reconstructive Surgery After Carcinological Excision
Keywords: Oral cancer; Free Flap; Neurrorhaphy; Quality of life
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Intervention Model Description: Comparison of primary and secondary outcomes measures between group 1 (resensitization by neurorrhaphy) and group 2 patients (No resensitization by neurorrhaphy).
  Patients randomly included in the groups according to a randomization software (RedCap)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resensitized group (Experimental): Patients with resensitized free flap by neurorrhaphy
  Interventions: Procedure: neurorrhaphy
- Non Resensitized group (Experimental): Patients without resensitized free flap by neurorrhaphy.
  Interventions: Procedure: neurorrhaphy

INTERVENTIONS:
Procedure: neurorrhaphy — During the surgery, the flap is removed from its donor site, placed on the recipient site (instead of carcinological excision) and its survival is ensured by arterial and venous anastomosis (to the artery and facial vein or to the external carotid artery and thyro-linguofacial veinous trunk).
  We then propose a reconstruction complement: nerve anastomosis (neurorrhaphy) to the lingual nerve for the antebrachioradial and anterolateral thigh flaps, and to the lower alveolar nerve for the fibular bone flaps. This supplement is performed during microsurgical time by a suture for the patient in group 1.

SUMMARY:
The surgical procedure consists in removing a tumor of the oral cavity and then repairing the oral defect by the use of a free flap. A free flap is tissue composed of skin and aponeurosis taken from the thigh or forearm, or tissue composed of bone taken from the leg to fill in tissue loss. This tissue is vascularized by a vein and an artery that are removed with the flap to ensure its survival. Investigator would also like to harvest the nerve involved in the sensitivity of the skin flap to suture it to a nerve which will be located near the reconstructed area, and this to enhance sensitivity of the reconstructed oral cavity. Thanks to this, investigator also wish to highlight that this resensitization would improve the patient's quality of life particularly regarding his major oral functions (swallowing, phonation, sensation of cold and hot felt, chewing).

Investigator therefore seek to demonstrate that suturing the nerve will give to the patient the ability back to feel tactile and thermal sensations This is the purpose of the study.

DETAILED DESCRIPTION:
Investigator will compare patients in whom the nervous suture will be performed and patients in whom it will not. If a significant difference in oral sensitivity is noted between these 2 groups, investigator can support our thesis: suturing the flap nerve increases its ability to regain sensitivity.

All patients are first diagnosed in consultation and presented at a carcinologic multidisciplinary consultation during which an individually adapted treatment is proposed (according to the French "Plan Cancer"). If it consists in a surgery with reconstruction using free flap technique at the same time, Investigator then propose to the patient to integrate our study. The possibility to participate to this study is therefore proposed to the patient on the same day that the plan of treatment is presented. The patient has a period of reflection, minimal time necessary to mature his reflection and make their choice with their loved ones and decide if they agree to participate to the study. His answer is required the day before the surgery. This represents a reflection period of two weeks on average. If he accepts it, computer software (RedCap®) will determine at random if the surgical team will perform a nervous suture or not. As a result, two groups patients are then created: one with nervous suture and one with no nervous suture. By comparing these two groups, investigator hope to demonstrate that there will be more patients with a flap sensitive in the "with nerve suture" group than in the "without nerve suture" group.

Investigator will then collect data from tests and questionnaires allowing us to judge the resensitization of the flap during follow-up consultations at 3, 6 months then at 1 year postoperatively in parallel follow-up consultations. That is to say that the patient therefore comes for a consultation as part of his cancer follow up and investigator take advantage of this time to carry out tests and questionnaires. This adds about 20 minutes of consultation time.

A preoperative evaluation will be done before the surgery corresponding to the basal state calibration. During these consultations, investigator perform two tests and investigator will provide 2 quality of life questionnaires to fill out:

* The two-discriminating points test: two points are applied on the flap at different distances and the patient must indicate if he feels one or two points.
* The hot/cold test: hot water and cold water are applied on the flap separately, and the patient should indicate if he feels the temperature differences.
* The QLQ-C30 and EOTRC H&N 35 questionnaires: several questions concerning the quality of life are asked to the patient who must answer them as honestly as possible.

After collecting all this information, investigator can compare the sensitivity of free flaps with or without nerve suture.

In parallel, investigator will also evaluate the economic impact and cost that this can represent by comparing the operating and hospitalization times of patients in each group. Investigator believe that the operating time is not increased nor the length of hospitalization and therefore that there is no additional cost.

ELIGIBILITY:
Inclusion Criteria:

* - Patient eligible for reconstructive surgery after carcinological excision following a decision taken in a multidisciplinary consultation, and for whom the envisaged oral defect concerns either the soft tissues of the oral cavity and oropharynx, or the mandibular bone
* Scheduled post-operative radiotherapy
* Coverage by the Social Security system
* Capacity to provide informed consent

Exclusion Criteria:

* Post-traumatic substance loss (ballistic autolysis)
* Surgical or anesthetic contraindication (physiological age, other proposed therapeutic options)
* Pregnant or breastfeeding woman
* Subject incapable of full age or deprived of liberty
* Indication for chemotherapy with highly neurotoxic agents
* Inability to complete questionnaires or express feelings during the examination
* Any situation judged by the investigator as a contraindication to neurorrhaphy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Epicritic sensitivity measurement | Before intervention (at day 1).
  It is a method of discriminating evaluation of epicritic sensitivity validated by the scientific literature
Thermoalgic sensitivity measurement | Before intervention (at day 1)
  Thermoalgic resensitization measured by Hot test
Thermoalgic sensitivity measurement | Before intervention (at day 1)
  Thermoalgic resensitization measured by cold test

SECONDARY OUTCOMES:
Quality of life judged by QLQ-C30 | Before intervention, 3 months post-surgery, 6 months post-surgery, 1 year post-surgery.
  The QLQ-C30 is a are self-administered questionnaire and validated by the European Organisation for Research and Treatment of Cancer assessing overall health status of patients. The QLQ-C30 focuses on patients' overall quality of life and disease experience
Quality of life judged by EOTRC H&N 35 | Before intervention, 3 months post-surgery, 6 months post-surgery, 1 year post-surgery.
  The EORTC H&N 35 questionnaires are self-administered and validated by the European Organisation for Research and Treatment of Cancer assessing overall health status of patients. The EORTC H&N 35 focuses on mouth sensations and major oral functions such as chewing, phonation or swallowing
Voice Handicap Index | Before intervention, 3 months post-surgery, 6 months post-surgery, 1 year post-surgery.
  The VHI is a self-assessment scale (established by Jacobson et al., 1997) adapted in French that provides a psychometric inventory of vocal disability that can be used for a wide variety of conditions (Woisard et al., 2004). The higher the score is, the greater the feeling of disability. The VHI is rated on 120 points. For each question, the scale used is a Likert analog scale, a frequency variable rated from 0 to 4 (0=never; 1=almost never; 2=sometimes; 3=almost always; 4=always). Its three subscales are each composed of 30 assertions
The Deglutition Handicap Index | 6 months post-surgery
  The DHI is a French self-administered questionnaire on the quality of life specific to swallowing. It was written and validated in 2006 by Woisard and Puech, based on the Voice Handicap Index (VHI) model (Crestani, Moerman et al.), (Woisard & Lepage, 2010). It consists of three domains, each containing ten items:
Economic evaluation | 1 month post-hospitalization
  The investigators collect the operating time and hospitalisation time for each patient to demonstrate that our operating technique does not generate any additional costs.
impact on the cost of the stay | 1 month post-hospitalization
  The investigators collect the operating time and hospitalisation time for each patient to demonstrate that our operating technique does not generate any additional costs.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud DEPEYRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France